CLINICAL TRIAL: NCT05870332
Title: Nationwide Study of Artificial Intelligence in Adenoma Detection for Colonoscopy
Acronym: NAIAD
Status: Recruiting | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: Medtronic (Industry); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 292323
Record Dates: First submitted 2023-05-02; First posted 2023-05-23 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Colonic Polyp; Colonic Adenoma; Colo-rectal Cancer
Keywords: Artificial Intelligence; Computer assisted detection (CADe); Colorectal cancer; Adenoma Detection Rate (ADR)
MeSH Terms: conditions — Colonic Polyps; Colonic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- All patients: Patient ≥18 years old, with capacity to consent, scheduled for diagnostic colonoscopy
  Interventions: Device: GI Genius (GIG)

INTERVENTIONS:
Device: GI Genius (GIG) — GIG is an artificial intelligence unit that assists human colonoscopist in real-time to detect polyps during colonoscopy.
  Four months collection period prior to activating GIG, then four months with GIG, and Four months afterwards without GIG
  Other Names: CADe

SUMMARY:
The goal of this trial is to determine whether use of a Computer Assisted Detection (CADe) programme leads to an increase in ADR for either units or individual colonoscopists, independent of setting or expertise

DETAILED DESCRIPTION:
This is a case-control study comparing adenoma detection rate (ADR) in hospitals (and individual colonoscopists), before, during and after use with an artificial intelligence unit called GI Genius™ (GIG). GIG is a Computer-assisted detection (CADe) module that assists the human colonoscopist in real-time, by detecting and marking out polyps during colonoscopy. It has been shown to be effective in expert colonoscopists, but the effect in non-expert, general, colonoscopists is not known.

The investigator wish to deploy GIG into colonoscopy through the UK using a step-wedge design. Sites will be randomly allocated a start date for GIG deployment, collecting data for four months prior to this. In this way, all sites will have the active intervention and will provide their own case-control data. (4 months collection prior to activating GIG, 4 months with GIG, 4 months afterwards without GIG)

The study will concentrate on non-expert colonoscopists, to determine whether GIG can increase ADR. Patients will undergo the same colonoscopy that they would have had in any case, with no additional trial visits or interventions. There will be no alteration to the usual care pathway from the patient's perspective.

If the investigator can prove GIG increases ADR in this way, it will provide support to roll out this technology routinely to improve the quality of colonoscopy nationwide.

ELIGIBILITY:
Inclusion Criteria:

* Any patient aged 18-85 scheduled for colonoscopy by current NHSE / British Society of Gastroenterology criteria

Exclusion Criteria:

* Colonoscopy being performed for polyp surveillance
* Unable to provide informed, written consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Unselected patients scheduled for diagnostic colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
CADe-ADR in real world practice | 24 months
  The primary outcome measure will be adenoma detection rate. This will be studied across three phases: prior to use of CADe (baseline practice), while using CADe (study period) and finally after CADe (without the device in situ: "washout" phase).

SECONDARY OUTCOMES:
APC | 24 months
  Mean adenomas per colonoscopy (APC)
Polyp characteristics | 24 months
  Polyp size (mm) and location (in colonic segments)
Procedure time | 24 months
  Total procedure (insertion+withdrawal) and withdrawal time

CONTACTS AND LOCATIONS:
Overall Officials: Prof Bu'Hussain B Hayee, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom